CLINICAL TRIAL: NCT04903795
Title: A Phase 1 Study of Bispecific T Cell Engager (BRiTE) in Patients With Newly Diagnosed or Recurrent Glioblastoma
Brief Title: BRiTE - Bispecific T Cell Engager for Patients With Glioblastoma
Acronym: BRiTE
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mustafa Khasraw, MBChB, MD, FRCP, FRACP (Other)
Collaborators: Adaptin Bio, Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Sponsor-Investigator, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108079
Record Dates: First submitted 2021-05-19; First posted 2021-05-27 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Newly Diagnosed Glioblastoma; Recurrent Glioblastoma
Keywords: EGFRvIII; Khasraw; BRiTE; Pro00108079
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- hEGFRvIII-CD3 (BRiTE) infusion (Experimental): Five escalating doses of continuously-infused BRiTE are planned: #1: 0.91 mcg/kg/day , #2: 2.88 mcg/kg/day, #3: 9.10 mcg/kg/day, #4: 28.78 mcg/kg/day, and #5: 91.00 mcg/kg/day.
  Interventions: Drug: hEGFRvIII-CD3 (BRiTE)

INTERVENTIONS:
Drug: hEGFRvIII-CD3 (BRiTE) — Bispecific T cell engager possessing one effector binding arm specific for the epsilon subunit of CD3 (a signaling molecule complex associated with the T cell receptor on T cells) while the opposing target-binding arm is directed against the hEGFRvIII epitope that is differentially expressed on the surface of tumor cells
  Other Names: BRiTE

SUMMARY:
This Phase 1 study will assess the safety of a novel brain Bispecific T cell engager (BRiTE) in patients with newly diagnosed or recurrent World Health Organization (WHO) Grade 4 glioblastoma (GBM). Owing to its short half-life, the study drug, BRiTE, will be continuously infused intravenously (IV) for 4 days (96 hours) in a 28-day cycle. Given that BRiTE specifically exerts its effects on tumor cells expressing the Epidermal Growth Factor Receptor variant III (EGFRvIII) mutation, we will only enroll patients with EGFRvIII-positive tumors in this study.

The primary objective is to evaluate the safety and tolerability of continually infused BRiTE in ndGBM and rGBM patients and determine the maximum tolerated dose (MTD) for continuously infused BRiTE.

DETAILED DESCRIPTION:
This proposed Phase 1 study will treat a maximum of 18 patients with pathologically documented supratentorial EGFRvIII-positive ndGBM or rGBM.

ndGBM patients: Participants with ndGBM must have undergone surgical resection of their tumor and completed standard of care RT with or without TMZ, depending on the status of O-6 methylguanine DNA methyltransferase (MGMT) promoter methylation as indicated below:

1) ndGBM patients with a methylated MGMT promoter should have received standard of care concomitant RT and TMZ, followed by 6 cycles of adjuvant TMZ, before they can participate in this study 2) ndGBM patients with an unmethylated MGMT promoter should have received standard of care RT, but need not have received concomitant TMZ or 6 cycles of adjuvant TMZ and can be enrolled 4 weeks after completion of standard of care RT 3) RT for 3 or 6-week courses are accepted as follows: i. Typically, 59.4-60 Gy over approximately 6 weeks duration, for patients under 65 years old ii. A minimum of 40 Gy over 3 weeks duration, for patients 65 years or older. Note: Patients who progress during RT or within 4 weeks after completion of RT are not eligible to participate in this study.

rGBM patients at first progression: Participants with rGBM can enroll if they have pathological or radiographic confirmation of their tumor recurrence. Patients that undergo total gross resection at time of recurrence are eligible to enroll.

Once deemed eligible upon screening, patients will receive a continuous IV infusion of BRiTE for 4 days (96 hours), followed by 24 days off-treatment, for a total period of 28 days. This 28-day period is 'Cycle 1'. Patients may continue receiving BRiTE infusions for 2 subsequent 'maintenance' cycles, each lasting for 28 days (Cycles 2 and 3): continuous BRiTE infusion for 4 days (96 hours), followed by 24 days off-treatment. Cohorts of 3 patients will be treated with increasing levels of continuously infused BRiTE in Cycle 1 to determine the MTD of BRiTE. Patients will be monitored for dose-limiting toxicity (DLT) during the DLT observation period that lasts for 28 days from the time of initiation of BRiTE infusion during Cycle 1. Patients will also be monitored for safety during the subsequent maintenance cycles of BRiTE. Along with safety, this study will include both preliminary assessments of clinical benefit and PK analysis of BRiTE.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old at the time of entry into the study
2. For both newly diagnosed and recurrent patients, pathologically documented supratentorial WHO grade 4 GBM with a confirmed EGFRvIII mutation at the most recent diagnosis, with radiographic contrast enhancing disease that is ≤ 4 cm in maximal diameter in any plane before resection.

   i. ndGBM patients: Must have undergone surgical resection of their tumor. Patients are still eligible if they have measurable or non-measurable residual enhancing tumor following resection, providing they meet all other eligibility criteria. Newly diagnosed patients must complete standard of care RT with or without TMZ before participation, depending on the MGMT promoter methylation status as follows:
   1. Patients with methylated MGMT promoter status should have received standard of care concomitant RT and TMZ, followed by 6 cycles of adjuvant TMZ, before they can participate in this study
   2. Patients with an unmethylated MGMT promoter status should have received standard of care RT, but need not have received concomitant TMZ or 6 cycles of adjuvant TMZ and can be enrolled after 4 weeks from completion of standard of care RT
   3. Patients whose MGMT status is unknown or indeterminate will be treated as though they have a methylated MGMT promotor status for eligibility purposes
   4. RT for 3 or 6-week courses are accepted as follows:

      * Typically, 59.4-60 Gy over approximately 6 weeks duration, if under 65 years old
      * A minimum of 40 Gy over 3 weeks duration, if 65 years or older
   5. Patients who progress during RT or within 4 weeks after completion of RT are not eligible.

   ii. rGBM patients at first progression: Must have pathological or radiographic confirmation of their tumor recurrence that is ≤ 4 cm in maximal diameter in any plane.

   Note: Patients that undergo total gross resection at time of recurrence are eligible to enroll. Patients are still eligible if they have measurable or non-measurable residual enhancing tumor following resection, providing they meet all other eligibility criteria.
3. Karnofsky Performance Score (KPS) ≥ 70%
4. Able to undergo brain MRI with and without contrast. Patients who cannot undergo MRI due to obesity or to having certain metal in their bodies (i.e. pacemakers, infusion pumps, metal aneurysm clips, metal prostheses, joints, rods, or plates) or patients with any known severe allergies to contrast agents are not eligible. Patients with mild allergies (i.e., rash only) are eligible for inclusion and can be pretreated with acetaminophen and diphenhydramine prior to injection of the contrast agent.
5. Hematological function as follows:

   i. Hemoglobin ≥ 9.0 g/dL ii. Absolute neutrophil count (ANC) ≥ 750/mm3 iii. Platelet count ≥ 50,000
6. Renal function as follows:

   i. Creatinine ≤ 1.5 x ULN
7. Hepatic function as follows:

   i. Aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN) ii. Alanine aminotransferase (ALT) ≤ 2.5 x ULN iii. Total bilirubin ≤ 1.5 x ULN Exception: Patient has known Gilbert's Syndrome or patient has suspected Gilbert's Syndrome, for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.
8. Patient or partner(s) meets one of the following criteria:

   1. Non-childbearing potential (i.e. not sexually active, physiologically incapable of becoming pregnant, including any person who is post-menopausal or surgically sterile, or any person who has had a vasectomy). Surgically sterile people are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Postmenopausal for purposes of this study is defined as 1 year without menses; or
   2. Childbearing potential and agrees to use one of the following methods of birth control: approved hormonal contraceptives (e.g. birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g. a condom or diaphragm) used with spermicide while on study and for an additional 4 months after completing the last infusion of BRiTE.
9. Patients of childbearing potential must have negative serum pregnancy test within 1 week of the 1st BRiTE infusion
10. A signed ICF approved by the IRB will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study

Exclusion Criteria for All Patients:

1. Patients who are pregnant or breastfeeding/chestfeeding
2. Patients with baseline corrected QT interval (QTc) > 480ms on screening electrocardiogram (ECG).

   Note: QTc measurements will use Fridericia's correction method (QTcF).
3. Known hypersensitivity to immunoglobulins or to any other component of BRiTE
4. Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate
5. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
6. Patients with severe, active co-morbidity, defined as follows:

   i. Patients with an active infection requiring IV treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C) ii. Patients with known immunosuppressive disease or known HIV infection, with CD4+ T cell counts < 350 cells/µl iii. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4) iv. Patients with known lung (forced expiratory volume in the first second of expiration [FEV1] < 50%) disease or uncontrolled diabetes mellitus v. Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy
7. Patients with known Human Immunodeficiency Virus (HIV) positive status only if CD4+ T cell counts < 350 cells/µl. Patients with known HIV and CD4+ T cell counts over 350 cells/µl are eligible.
8. Patients with known hepatitis C virus (HCV) positive status, who have not completed curative antiviral treatment and have HCV viral load above the limit of quantification. Patients with well-controlled HCV are eligible.
9. Patients with known hepatitis B virus (HBV) infection, with evidence of a hepatitis B surface antigen, indicative of an active infection. Patients with well-controlled HBV are eligible.
10. Patients on corticosteroids ≥ 2 mg dexamethasone daily or equivalent within 7 days of 1st BRiTE infusion
11. Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months
12. Toxicities from prior antitumor therapy that have not resolved to CTCAE version 5.0 grade 1 (with the exception of AEs reflecting myelosuppression such as neutropenia, anemia, or thrombocytopenia), or to levels dictated in the eligibility criteria. Other exceptions include alopecia or toxicities from prior antitumor therapy that are considered irreversible (defined as having been present and stable for > 2 months) are allowed if they are not otherwise described in the exclusion criteria.

Exclusion Criteria for ndGBM Patients Only:

1. Patients who previously received other therapeutic interventions for ndGBM, with the exception of surgical resection and standard of care concomitant RT and TMZ (including adjuvant TMZ) for their brain tumor
2. Patients who have had only a biopsy prior to receiving standard of care concomitant RT and TMZ
3. Unmethylated MGMT patients who have received RT < 4 weeks prior to initiation of BRiTE infusion

Exclusion Criteria for rGBM Patients Only:

1. Patients who have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks), or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to enrollment unless patients have recovered from side effects of such therapy
2. Patients who have received immunotherapy prior to enrollment
3. Patients less than 12 weeks from RT, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Begins with the infusion of BRiTE during Cycle 1 and goes through 28 days from the time of initiation of the infusion
  Proportion of patients with DLT within each dose level

SECONDARY OUTCOMES:
Objective response rate (ORR) | 8 weeks
  ORR per Response Assessment in Neuro-Oncology Criteria (RANO 2.0)
Pharmacokinetic (PK) of BRiTE observed during Cycle 1 of BRiTE infusion | Prior to initiation of Cycle 1 (each cycle is 28 days) of BRiTE infusion (baseline; on Day 0) till 1 hour after the end of infusion (on Day 4)
  Changes in levels of BRiTE from baseline (prior to start of BRiTE infusion)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — https://www.dukehealth.org/clinical-trials